CLINICAL TRIAL: NCT00426712
Title: A Phase 1, Randomized, Observer-blind, Dose-escalating Study in Adult End-stage Renal Failure Patients to Explore the Safety, Tolerability, Pharmacokinetics and Immune Response to Recombinant Hepatitis B Virus Surface Antigen (rHBsAg) Co-administered With Dynavax Immunostimulatory Phosphorothioate Oligodeoxyribonucleotide (1018 ISS)
Brief Title: Safety of HEPLISAV™ Hepatitis B Virus Vaccine in End-stage Kidney Failure Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DV2-HBV-09
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis B
Keywords: Chronic kidney failure; Chronic kidney disease; Hemodialysis; HBV vaccine; Hepatitis B vaccine; Hepatitis B; Hepatitis; HBV; Prevention & Control
MeSH Terms: conditions — Hepatitis B; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Hepatitis | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Low dose
  Interventions: Biological: 1018 ISS immunostimulatory oligonucleotide with HBV surface antigen
- 2 (Experimental): Middle dose
  Interventions: Biological: 1018 ISS immunostimulatory oligonucleotide with HBV surface antigen
- 3 (Experimental): High dose
  Interventions: Biological: 1018 ISS immunostimulatory oligonucleotide with HBV surface antigen
- 4 (Active Comparator)
  Interventions: Biological: Hepatitis B Vaccine (Recombinant)

INTERVENTIONS:
Biological: 1018 ISS immunostimulatory oligonucleotide with HBV surface antigen — Intramuscular (IM) injections on Day 0, Week 4 and Week 24, plus a placebo (salt solution) injection at Week 8
  Other Names: HEPLISAV™
  Arms: 1; 2; 3
Biological: Hepatitis B Vaccine (Recombinant) — IM (in the muscle) injections on Day 0, Week 4, Week 8 and Week 24
  Other Names: ENGERIX-B®
  Arms: 4

SUMMARY:
The purpose of this study is to find out if a new investigational hepatitis B virus vaccine, HEPLISAV™, is safe in patients at least 40 years of age who have progressive loss of kidney function with more advanced stage 3 (GFR ≤ 45 mL/min) or stage 4 chronic kidney disease, and are expected to eventually go on hemodialysis.

DETAILED DESCRIPTION:
Infection with hepatitis B virus (HBV) is a major global health problem. Worldwide, it is estimated that 2 billion people have been infected previously and 350 million are chronically infected. About 25% of people who do not initially clear the infection will later develop chronic active hepatitis. Hemodialysis and pre-dialysis patients with kidney failure have multiple immune defects that make them more likely to develop a chronic infection. In addition, hemodialysis increases the risk of exposure to HBV. Existing HBV vaccines are effective in preventing infection in healthy adults. However, poor responses occur in people who are over 40 years of age and have end-stage kidney failure.

This study will evaluate the safety, tolerability and immune response of three escalating dose levels of HEPLISAV™, compared with a commercially available HBV vaccine, Engerix-B®, in patients at least 40 years of age who have progressive loss of kidney function with more advanced stage 3 (GFR ≤ 45 mL/min) or stage 4 chronic kidney disease and are expected to eventually go on hemodialysis. About 72 patients will be included in the study. Once patients have been consented, screened, and randomized to treatment, they will receive four injections over a 24-week period, with follow-up visits at 28 and 50 weeks. Safety and tolerability will be evaluated by occurrence of adverse events, periodic laboratory tests, vital signs, and local/systemic reactogenicity.

Comparison: Patients will receive treatment with one of three escalating dose levels of HEPLISAV™ or the comparator vaccine, Engerix-B®.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Progressive loss of kidney function with more advanced stage 3 (GFR at least 45 mL/min) or stage 4 chronic kidney disease by National Kidney Foundation classification, and are expected to eventually go on hemodialysis
* Body mass index of 31 or less

Exclusion Criteria:

* Received previous vaccination with any HBV vaccine (1 or more doses)
* Any history of HBV infection
* Pregnant or breast-feeding, or planning a pregnancy during the study
* Has autoimmune disease
* Diagnosis of chronic kidney failure due to autoimmune disease
* Receiving hemodialysis treatment at the time of enrollment
* Received any blood products or antibodies within 3 months prior to study entry, or is likely to require blood products during the study
* Ever received an injection with DNA plasmids or oligonucleotides
* Received erythropoietin within 7 days prior to the first study injection
* Received vaccination with any vaccines during the 4 weeks prior to study entry
* Received any other investigational medicinal agent during the 4 weeks prior to study entry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events and local and systemic reaction rates | 28 weeks

SECONDARY OUTCOMES:
Portion of subjects who have a seroprotective immune response (anti-HBsAg antibody ≥ 10 mIU/mL) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, DPhil, Study Director — Dynavax Technologies Corporation
Locations (4):
- United States (4):
  - West Coast Clinical Trials, Costa Mesa, California
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Covance, Austin, Texas
  - University of Virginia Health System, Nephrology Clinical Research Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
3/2017 No change to status of this study

REFERENCES:
- See also: Dynavax Webpage — http://www.dynavax.com